CLINICAL TRIAL: NCT07145866
Title: Evaluation of Varenicline and Accelerated TMS for Reduction of Nicotine Use
Brief Title: Varenicline and Accelerated Transcranial Magnetic Stimulation (TMS) for Quitting Nicotine Use (Pilot Study)
Acronym: V-TMS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jodi Gilman, Associate Professor, Harvard Medical School; Director of Neuroscience, Center for Addiction Medicine, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P001964
Record Dates: First submitted 2025-08-12; First posted 2025-08-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Nicotine Dependence; Transcranial Magnetic Stimulation; Vaping; Smoking Cessation; Smoking (Tobacco) Addiction
Keywords: Vaping; Smoking; Nicotine; Adults; Cessation; Varenicline; Transcranial Magnetic Stimulation; TMS
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Smoking Cessation; Smoking; Behavior, Addictive | interventions — Varenicline; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Up to 90 participants will be consented, and approximately 30 participants will be randomized in a double-blind, 2-arm parallel design clinical trial comparing nicotine use abstinence rates in participants randomly assigned to: 1) varenicline + active TMS, or 2) varenicline + sham TMS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Varenicline + Active TMS (Active Comparator): In this arm, participants will take 12 weeks of varenicline. They will also receive 5 consecutive days of 5 hourly TMS treatments, adjusted to an individualized target specific to the participant based on their brain MRI collected at the baseline imaging visit. Participants will also receive 6 brief nicotine cessation counseling sessions.
  Interventions: Drug: varenicline; Device: Transcranial Magnetic Stimulation; Behavioral: Nicotine Cessation Counseling
- Varenicine + Sham TMS (Sham Comparator): In this arm, participants will receive 12 weeks of varenicline and instructions on how to take it. They will also receive 5 consecutive days of 5 hourly TMS treatments, adjusted to an individualized target specific to the participant based on their brain MRI collected at the baseline imaging visit. However, the sham setting will deliver no magnetic field to the brain; instead, it will deliver electrical current to the scalp to mimic the feel of active treatment. Participants will also receive 6 brief nicotine cessation counseling sessions.
  Interventions: Drug: varenicline; Device: Transcranial Magnetic Stimulation Sham; Behavioral: Nicotine Cessation Counseling

INTERVENTIONS:
Drug: varenicline — Dosing of this FDA-approved medication will follow the below schedule, which follows the clinical standard:
  0.5 mg once daily or 3 days, 0.5 mg twice daily for 4 days 1.0 mg twice daily for 11 weeks
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a noninvasive FDA-approved technique that is commonly used as a treatment for depression and has been approved for use in smoking cessation. In this study, TMS will be administered within FDA-approved guidelines under the supervision of a physician with experience in administering the treatment and monitoring for complications. Following an accelerated model, it will consist of 5 hourly treatments for 5 consecutive days.
  Arms: Varenicline + Active TMS
Device: Transcranial Magnetic Stimulation Sham — Transcranial magnetic stimulation (TMS) is a noninvasive FDA-approved technique that is commonly used as a treatment for depression and has been approved for use in smoking cessation. In this study, TMS will be administered within FDA-approved guidelines under the supervision of a physician with experience in administering the treatment and monitoring for complications. Following an accelerated model, it will consist of 5 hourly treatments for 5 consecutive days. The sham setting will deliver no magnetic field to the brain but will deliver electrical current to the scalp to mimic the feel of active treatment.
  Arms: Varenicine + Sham TMS
Behavioral: Nicotine Cessation Counseling — Each participant will receive 6 sessions of brief nicotine cessation counseling by a trained study staff member. This will be provided at the weekly follow-up visits, spread out throughout the study. This counseling, while not the main aim of the study, should help participants manage their expectations of quitting and provide support and quitting strategies throughout the process.

SUMMARY:
The goal of this clinical trial is to learn if a combination of varenicline and accelerated Transcranial Magnetic Stimulation (aTMS) works to help adults quit using nicotine products. Researchers will compare varenicline + active aTMS to varenicline + sham (inactive) aTMS to see the effect of aTMS on reaching abstinence. The main question it aims to answer is: Does receiving active aTMS + varenicline lead to higher abstinence rates and lower nicotine craving?

Participants will be asked to:

* Complete 2 brain MRI scans
* Take varenicline every day for 12 weeks
* Quit using nicotine products at the end of the second week of varenicline
* Complete 5 consecutive days (Monday-Friday, uninterrupted) of TMS treatments
* Complete 12 brief, weekly follow-up visits
* Complete a brief daily survey each day that they take the study drug

DETAILED DESCRIPTION:
This is a 12-week randomized parallel design, double-blind, 2-arm clinical trial consisting of a combination of circuit-targeted TMS and varenicline in 30 adults aged 18-65 with nicotine use disorder who would like to reduce or stop nicotine use.

Eligible participants will complete a baseline assessment of questionnaires and laboratory assessments. They will be randomized to receive varenicline and either active or sham TMS. Participants will be randomized at their baseline scan visit, during which they will undergo urinalysis, an fMRI scan, and a task and questionnaire battery. At this visit, participants will receive the study medication and will be instructed to take it for 12 weeks titrated to 1mg twice daily over seven days.

Shortly after, participants will complete a TMS treatment preparation visit during which the treatment target is located and stimulation intensity of the TMS is determined. This target is used in the subsequent TMS Treatment Week consisting of 5 consecutive days of 5 TMS treatments per day. Participants' quit date will be set for the Saturday following their TMS treatments. The week after completing their TMS treatments, they will return for a second imaging visit identical to the baseline scan.

Each week of the varenicline treatment period, participants will complete weekly follow-ups with study staff, either virtually or in-person, to determine nicotine use and complete questionnaires regarding their substance use in the past week, depression, and anxiety. Six of these visits will include brief sessions of nicotine use cessation counseling with a trained study staff member.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤65;
* The ability to give written, informed consent;
* Fluency in English;
* Reported interest in quitting nicotine vaping or smoking within the next month;
* Nicotine dependence, as defined by a score of ≥4 on the 10-question E-cigarette Dependence Inventory (ECDI) or Fagerström Test for Nicotine Dependence (FTND);
* Smoke or vape nicotine daily for at least the past 90 days, as confirmed by self-report and timeline follow-back methods;
* Saliva cotinine >30ng/mL;

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Use of smoking cessation pharmacotherapy in the past month;
* Unwilling to abstain during the study from using smoking cessation aids other than those provided by the study;
* Prior adverse drug reaction to varenicline;
* Receiving or planning to receive other TMS treatments or investigational drugs during course of participation
* Contraindications to TMS (including seizures, metallic implants, severe existing tinnitus, etc.);
* Contraindications to MRI (including presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia);
* Inpatient psychiatric hospitalization or suicide attempts in the past six months, or recent active suicidal ideation or suicidal behavior identified at enrollment or baseline visits;
* History of seizures and/or history of TBI subtypes associated with elevated seizure risk (e.g. penetrating injury and intraparenchymal hemorrhage)
* History of unstable neurological illness or major medical illness, such as epilepsy or renal impairment, in the past six months, unless clearly resolved;
* In the opinion of the investigators, evidence of active problem substance use severe enough to compromise ability to safely participate;
* In the opinion of the investigators, unable to safely participate in this study and/or provide reliable data (e.g., claustrophobia, unable to tolerate TMS or MRI procedures, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Biochemically-confirmed continuous nicotine abstinence across study weeks 9-12 | Week 9-Week 12
  Point-prevalence abstinence from e-cigarette use was defined as self-report of no e-cigarette use since the last visit, bioverified by saliva cotinine <30 ng/ml. Continuous abstinence is defined as observed point-prevalence abstinence over specified study visits at weeks 9, 10, 11 and 12. The primary analysis will compare the proportion of participants achieving continuous abstinence in the TMS + varenicline group versus the Sham + varenicline group using a chi-square test. If expected cell counts are low (<5 in any cell), Fisher's exact test will be used instead.
Resting State Functional Connectivity (rsFC) | Baseline, Week 12
  Within-network resting state Functional Connectivity (rsFC) will be computed by extracting the mean BOLD time series from each region of interest comprising the addiction circuit and calculating pairwise Pearson correlations, which will then be Fisher z-transformed and averaged across all ROI pairs to derive a single within-network rsFC metric per participant at each time point. To isolate effects at the circuit level rather than changes induced by stimulation of the medial prefrontal cortex (mPFC) target site itself, the mPFC stimulation region will be excluded from the connectivity analyses. The primary analytic approach will use a linear mixed-effects model with fixed effects for time (baseline vs. post-treatment), treatment group (TMS vs. sham TMS), and their interaction, as well as a random intercept for each participant.
Change in Insula Activation to Nicotine Cues During a Cue Reactivity Task Measured by fMRI | Baseline, Week 12
  Neural responses to nicotine and neutral cues will be modeled, convolved with the canonical hemodynamic response function, and contrast images for nicotine > neutral cues will be generated for each participant at each time point. These contrast images will be entered into second-level analyses to test group-level effects. The primary region of interest (ROI) will be the bilateral anterior insula, defined using an anatomical mask from the Harvard-Oxford atlas. The main analytic model will be a mixed-effects repeated-measures ANOVA or linear mixed-effects model with fixed effects of time (pre vs. post), treatment group (TMS + varenicline vs. sham TMS + varenicline), and their interaction, with subject-level random intercepts. The key test of our hypothesis is the time × treatment interaction within the anterior insula ROI, which reflects whether treatment modulates cue-elicited insula activity.

SECONDARY OUTCOMES:
7-day point prevalence abstinence at Week 12 | Week 12
  Point-prevalence abstinence from e-cigarette use was defined as self-report of no e-cigarette use since the last visit, bioverified by saliva cotinine <30 ng/ml.
Nicotine withdrawal symptoms | Baseline, Week 12
  Minnesota Nicotine Withdrawal Scale (MNWS) total scores over study weeks 1 to 12. The MNWS is an 8-item measure assessing the severity of nicotine withdrawal symptoms. Items are scored on an ordinal scale from 0 ("not at all") to 4 ("extreme") with total scores ranging from 0 to 32. Higher scores indicate greater severity of nicotine withdrawal symptoms.
Nicotine Craving (vaping) | Baseline, Week 12
  Summed scores from the Questionnaire of Vaping Craving (QVC) over Study Weeks 1 to 12. The QVC is a 10-item self-rated validated measure (ranging from 10 to 70) of vaping craving that examines desire and intent to vape and anticipation of positive outcomes related to e-cigarette use, with higher scores indicating greater cravings to vape. This is applicable to those who report using e-cigarettes.
Nicotine Craving (smoking) | Baseline, Week 12
  Summed scores from the Questionnaire on Smoking Urges-Brief (QSU-Brief) over Study Weeks 1 to 12. This is a 10-item self-report measure of smoking urges and cravings with scores ranging from 10-70; higher scores indicate greater cravings to smoke. This is applicable to those who report smoking cigarettes.
Change in Depressive Symptoms | Baseline, Week 12
  The Beck Depression Inventory-II (BDI-II) will be used to assess symptoms of depression. The scale ranges from 0 - 63, with a higher score indicating greater depression.
Change in Anxiety Symptoms | Baseline, Week 12
  The Beck Anxiety Inventory (BAI) will be used to assess the frequency of anxiety symptoms, including cognitive and somatic symptoms. Higher scores indicate greater anxiety severity, with scores ranging from 0-63.

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events during the treatment period [Safety] | Week 0-Week 12
  Open-ended questioning will be used to assess adverse events throughout the trial. This outcome reports on the number of participants who reported at least one adverse event between the first imaging visit (Week 0) to the end of treatment (Week 12).

CONTACTS AND LOCATIONS:
Overall Officials: Jodi M Gilman, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No